CLINICAL TRIAL: NCT00052884
Title: A Phase I Study of Amifostine Followed by High-Dose Escalation of Melphalan With Stem Cell Reconstitution for Patients With Primary Systemic Amyloidosis
Brief Title: Amifostine and Melphalan in Treating Patients With Primary Systemic Amyloidosis Who Are Undergoing Peripheral Stem Cell Transplantation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual and changes in clinical practice
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258785; U10CA021115 (NIH); ECOG-E2A01
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: drug/agent toxicity by tissue/organ; primary systemic amyloidosis
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Amifostine; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amifostine, Melphalan, and Stem Cell Reconstitution (Experimental): Amifostine, Melphalan, and Stem Cell Reconstitution. Doses of Melphalan tested included 100 mg/m2 and 120 mg/m2
  Interventions: Biological: filgrastim; Drug: amifostine trihydrate; Drug: melphalan; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: amifostine trihydrate
Drug: melphalan
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of plasma cells, either by killing the cells or by stopping them from dividing. Having a peripheral stem cell transplant to replace the blood-forming cells destroyed by chemotherapy, allows higher dose of chemotherapy to be given so that more plasma cells are killed. Giving a chemoprotective drug such as amifostine may protect kidney cells from the side effects of chemotherapy.

PURPOSE: This phase I trial is studying the side effects and best dose of melphalan given together with amifostine in treating patients who are undergoing peripheral stem cell transplant for primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of high-dose melphalan administered with amifostine in patients with primary systemic amyloidosis undergoing autologous peripheral blood stem cell transplantation.
* Determine the toxicity of high-dose melphalan when administered at the MTD in these patients.
* Determine the response rate in patients treated with this regimen.

OUTLINE: This is a nonrandomized, multicenter, dose-escalation study of melphalan.

Patients receive filgrastim (G-CSF) subcutaneously once daily until peripheral blood stem cell (PBSC) collection is complete. Apheresis begins on day 5 of G-CSF administration and continues until the target number of PBSCs are collected.

Within 6 weeks of PBSC collection, patients receive amifostine IV over 5 minutes on days -2 and -1 and high-dose melphalan IV over 30-60 minutes on day -1. Patients undergo autologous PBSC infusion on day 0.

Cohorts of 3-6 patients receive escalating doses of melphalan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 10 patients are treated at that dose.

Patients are followed approximately 3 months following transplantation, then every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 3-46 patients will be accrued for this study within 2.3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed amyloidosis

  * No secondary familial or localized amyloidosis
* Presence of monoclonal protein by immunoelectrophoresis or immunofixation of serum or urine
* No primary amyloidosis manifested only by carpal tunnel syndrome or purpura
* Amyloid deposits in a plasmacytoma or in bone marrow vessels in an asymptomatic individual not considered an amyloid syndrome

  * Amyloid syndromes include any of the following:

    * Hepatomegaly
    * Cardiomyopathy
    * Nephrotic range proteinuria
    * Peripheral or autonomic neuropathy
* No multiple myeloma defined by 1 of the following:

  * Presence of lytic bone disease
  * More than 30% bone marrow plasma cells

PATIENT CHARACTERISTICS:

Age

* 18 to 70

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Platelet count at least 100,000/mm^3

Hepatic

* See Disease Characteristics
* Total or direct bilirubin no greater than 2.0 mg/dL
* Alkaline phosphatase no greater than 4 times upper limit of normal

Renal

* See Disease Characteristics
* Creatinine less than 3.0 mg/dL

Cardiovascular

* See Disease Characteristics
* Ejection fraction at least 45% by echocardiogram
* No New York Heart Association class III or IV heart disease
* Systolic blood pressure ≥ 90 mmHg

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* No other malignancy within the past 5 years except surgically treated carcinoma in situ of the cervix, nonmelanoma skin cancer, or indolent prostate cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior interferon

Chemotherapy

* At least 4 weeks since prior melphalan
* Lifetime total melphalan dose less than 150 mg/m^2 (based on ideal body weight)

Endocrine therapy

* At least 4 weeks since prior dexamethasone

Radiotherapy

* No prior radiotherapy for amyloidosis

Surgery

* Not specified

Other

* No antihypertensive medications for at least 24 hours prior to, during, and for 1 hour after amifostine administration
* No other prior treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-01-22 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Assessed over 30 days
  The maximum tolerated dose is the highest dose level at which fewer than 1 of 3 or 2 of 6 patients experience dose-limiting toxicity, defined as any grade 3 or higher toxicity of any of the following: renal failure, alkaline phosphatase elevation, GI bleeding, and cardiac rhythm disturbances, assessed using NCI Common Toxicity Criteria, version 2.0.

CONTACTS AND LOCATIONS:
Overall Officials: Morie A. Gertz, MD, Study Chair — Mayo Clinic
Locations (16):
- United States (16):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Case Comprehensive Cancer Center, Cleveland, Ohio